CLINICAL TRIAL: NCT07332156
Title: Lung Cancer Incidence in Patients With Type 2 Diabetes and COPD: A Real-World Retrospective Cohort Study Comparing SGLT2 Inhibitors and Sulfonylureas
Brief Title: Lung Cancer Risk in Type 2 Diabetes With COPD: SGLT2 Inhibitors vs. Sulfonylureas
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Danbee Kang, Associate Professor, Samsung Medical Center
Other Study IDs: SU vs. SGLT2 in T2DM with COPD
Record Dates: First submitted 2025-12-28; First posted 2026-01-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; COPD (Chronic Obstructive Pulmonary Disease); Lung Cancer (Diagnosis)
Keywords: SGLT2 inhibitor; Sulfonylurea; T2DM with COPD; Lung cancer
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pulmonary Disease, Chronic Obstructive; Lung Neoplasms; Disease | interventions — Sodium-Glucose Transporter 2 Inhibitors; Sulfonylurea Compounds; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Treatment group (main): Users of SGLT2 inhibitors (for ITT analysis)
  Interventions: Drug: SGLT2 inhibitor
- Active control group (main): Users of sulfonylureas for ITT analysis
  Interventions: Drug: Sulfonylureas (SU)
- Treatment group (S1): Users of SGLT2 inhibitors (for ITT analysis)
  Interventions: Drug: SGLT2 inhibitor
- Active control group (S1): Users of DPP4 inhibitors (for ITT analysis)
  Interventions: Drug: Sulfonylureas (SU)
- Treatment group (S2): Users of SGLT2 inhibitors (for as-treated analysis)
  Interventions: Drug: SGLT2 inhibitor
- Active control group (S2): Users of sulfonylureas (for as-treated analysis)
  Interventions: Drug: DPP4 inhibitors

INTERVENTIONS:
Drug: SGLT2 inhibitor — Any new prescription of SGLT2 inhibitors after new onset of T2DM
  Groups: Treatment group (S1); Treatment group (S2); Treatment group (main)
Drug: Sulfonylureas (SU) — Any new prescription of sulfonylureas after new onset of T2DM
  Groups: Active control group (S1); Active control group (main)
Drug: DPP4 inhibitors — Any new prescription of DPP4 inhibitors after new onset of T2DM
  Groups: Active control group (S2)

SUMMARY:
The goal of this observational study is to learn if a specific diabetes medicine can lower the risk of lung cancer in people with type 2 diabetes and chronic obstructive pulmonary disease (COPD).

The main question it aims to answer is:

- Does taking medicines called SGLT2 inhibitors lower the chance of getting lung cancer compared to medicines called sulfonylureas?

Researchers will compare the medical records of people taking SGLT2 inhibitors to those taking sulfonylureas to see if the SGLT2 group has fewer cases of lung cancer.

Participants will not need to visit a doctor or take new medicines for this study. Researchers will use information from existing medical records to answer the research question.

DETAILED DESCRIPTION:
Study Design: This is a comparative effectiveness research study utilizing large-scale, population-based Real-World Data (RWD). By analyzing longitudinal data from existing medical records, researchers will emulate a target trial to minimize bias and provide robust estimates of the treatment effect.

Statistical Analysis Plan: The study employs a rigorous analytic framework consisting of a primary analysis and multiple sensitivity analyses to ensure the validity of the findings:

Primary Analysis: A comparison of SGLT2 inhibitors versus sulfonylureas using an Intention-To-Treat (ITT) framework, with follow-up censored upon treatment switching to estimate the effect of the initial treatment choice.

Sensitivity Analysis 1 (Active Comparator): A comparison of DPP-4 inhibitors versus SGLT2 inhibitors using the same ITT framework (censoring on switching) to assess the consistency of the results against an alternative second-line antidiabetic class.

Sensitivity Analysis 2 (As-Treated): A comparison of SGLT2 inhibitors versus sulfonylureas using an As-Treated approach, defining continuous use with a permissible gap (grace period) of 60 days between prescriptions to account for adherence patterns.

Significance and Impact Current guidelines for diabetes management prioritize cardiovascular and renal protection. This study aims to expand the clinical evidence base by:

* Providing actionable Real-World Evidence (RWE) on the long-term cancer-related outcomes of diabetes medications.
* Evaluating whether the choice of antidiabetic agents can serve as a strategy for lung cancer prevention in high-risk groups (COPD-T2DM).
* Contributing to the development of comprehensive treatment guidelines that consider cancer prevention alongside metabolic, cardiac, and renal health.

Abbreviation:

COPD, Chronic Obstructive Pulmonary Disease; DPP-4, Dipeptidyl Peptidase-4; ICD-10, International Classification of Diseases, 10th Revision; ICS, Inhaled Corticosteroids; ITT, Intention-To-Treat; LABA, Long-Acting Beta-2 Agonists; LAMA, Long-Acting Muscarinic Antagonists; RWD, Real-World Data; RWE, Real-World Evidence; SABA, Short-Acting Beta-2 Agonists; SAMA, Short-Acting Muscarinic Antagonists; SGLT2, Sodium-Glucose Cotransporter-2; SU, Sulfonylurea; T2DM, Type 2 Diabetes Mellitus;

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥40 years with prior COPD (from 2009) and newly diagnosed diabetes who initiated SU or SGLT2i between January 1, 2014 and December 31, 2023

Exclusion Criteria:

* Pre-existing
* ESRD
* Cancer
* Concurrent prescribing of the study drugs at the index date
* Exposure to the drugs of interest during the year preceding the index date
* Death or cancer incidence within a month

In the sensitivity analysis, we are planning to substitute sulfonylurea to DPP4 inhibitors.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included adults aged ≥40 years with a prior history of COPD (screened from 2009) and newly diagnosed type 2 diabetes who initiated treatment with either sulfonylureas or SGLT2 inhibitors between January 1, 2014, and December 31, 2023. Type 2 diabetes was defined as having two or more diagnosis records within one year using ICD-10 codes E10-E14. COPD was defined by the presence of ICD-10 codes J43 or J44 (excluding J43.0) concurrent with the prescription of COPD medications at least twice within a year; these medications included long-acting muscarinic antagonists (LAMA), long-acting beta-2 agonists (LABA), ICS plus LABA, short-acting muscarinic antagonists (SAMA), short-acting beta-2 agonists (SABA), SAMA plus SABA, methylxanthines, and systemic beta agonists.
  In the sensitivity analysis, we are planning to substitute sulfonylurea to DPP4 inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 21692 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Lung cancer | From index date + 30 days to the end of follow-up
  ICD-10 code (C33 or C34) and code for special purposes (V193)

SECONDARY OUTCOMES:
COPD exacerbation | From index date + 30 days to the end of follow-up
  COPD (J43 or J44, not J43.0) and antibiotics or steroids prescription and (emergency department or admission)
Any cancer | From index date + 30 days to the end of follow-up
  ICD-10 code ('C' code) and code for special purposes (V193)

IPD SHARING:
Plan to Share IPD: No